CLINICAL TRIAL: NCT06862388
Title: Clinical Research on Umbilical Cord Mesenchymal Stem Cells Therapy for Patients with Subacute Intracerebral Hemorrhage
Brief Title: Stem Cell Therapy for Intracerebral Hemorrhage
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang Zhouping (Other)
Collaborators: Wuhan Hamilton Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Tang Zhouping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202502088; ChiCTR2500095990 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2023-11-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Intracerebral Hemorrhage; Mesenchymal Stem Cell
Keywords: Intracerebral hemorrhage; Human umbilical cord mesenchymal stem cells; Stem cell therapy; Inflammation; Neural repair
MeSH Terms: conditions — Cerebral Hemorrhage; Inflammation | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: The clinical trial was divided into phase I and Phase II. The Phase I clinical trial is a Sequential design, and the Phase II clinical trial is a Parallel design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PhaseⅠclinical trial: 3+3 dose-escalation design (Experimental): The Phase I clinical trial is a 3+3 dose-escalation trial, with three dose groups, each including at least 3 subjects. The trial begins with the low-dose group. If the dose-limiting toxicity (DLT) assessment during the observation period meets the criteria of the 3+3 dose-escalation design, enrollment will proceed to the next higher dose group. Each subject will receive one dose of human umbilical cord mesenchymal stem cells (UC-MSCs) therapy, in addition to the standard treatment for intracerebral hemorrhage.
  Interventions: Biological: Device: Phase Ⅰ Dose Level 1; Biological: Device: Phase Ⅰ Dose Level 2; Biological: Device: Phase Ⅰ Dose Level 3
- Phase Ⅱ clinical trial: MTD group (Experimental): The Phase II clinical trial included two groups. The dose of UC-MSCs received in each group patients will be determined based on the phase I results. One of the two groups subjects received the MTD obtained in phase I, and the other group subjects received a dose lower than the MTD. Each subject in the Phase II clinical trial received three dose of stem cell therapies after enrollment.The second therapy is 7 days after the first therapy, and the third therapy is 7 days after the second therapy.
  Interventions: Biological: Device: Phase II MTD in Phase I
- Phase Ⅱ clinical trial: lower than the MTD group (Experimental): The Phase II clinical trial included two groups. The dose of UC-MSCs received in each group patients will be determined based on the phase I results. One of the two groups subjects received the MTD obtained in phase I, and the other group subjects received a dose lower than the MTD. Each subject in the Phase II clinical trial received three dose of stem cell therapies after enrollment.The second therapy is 7 days after the first therapy, and the third therapy is 7 days after the second therapy.
  Interventions: Biological: Device: Phase II lower than the MTD in Phase I

INTERVENTIONS:
Biological: Device: Phase Ⅰ Dose Level 1 — Patients in the first dose level will receive a cell dose of 1×10^6 cells/kg.
  Arms: PhaseⅠclinical trial: 3+3 dose-escalation design
Biological: Device: Phase Ⅰ Dose Level 2 — Patients in the second dose level will receive a cell dose of 2×10^6 cells/kg.
  Arms: PhaseⅠclinical trial: 3+3 dose-escalation design
Biological: Device: Phase Ⅰ Dose Level 3 — Patients in the third dose level will receive a cell dose of 4×10^6 cells/kg. Based on these findings, the maximum tolerated dose (MTD) will be determined.
  Arms: PhaseⅠclinical trial: 3+3 dose-escalation design
Biological: Device: Phase II MTD in Phase I — This group subjects received the MTD obtained in phase I.
  Arms: Phase Ⅱ clinical trial: MTD group
Biological: Device: Phase II lower than the MTD in Phase I — This group subjects received a dose lower than the MTD
  Arms: Phase Ⅱ clinical trial: lower than the MTD group

SUMMARY:
Intracerebral hemorrhage (ICH) is a common condition with high morbidity, mortality, and disability. The current treatments for ICH primarily include surgical and pharmacological interventions. For large hematomas, surgical options such as craniotomy, debridement, decompression, and minimally invasive hematoma aspiration may be performed. Pharmacological treatments are mainly symptomatic. Despite timely and standardized surgical or pharmacological interventions, many patients with ICH still experience significant sequelae, which severely affect their quality of life and place a substantial burden on both families and society. Currently, there are limited drugs available specifically for the treatment of ICH.

In recent years, stem cell therapy has gained attention as a promising treatment for neurological diseases. Human umbilical cord mesenchymal stem cells (UC-MSCs) are multifunctional stem cells with properties such as self-renewal, multidirectional differentiation potential, tissue repair, immunomodulation, and anti-inflammatory effects. Studies have shown that intravenous transplantation of UC-MSCs is safe, and their application in the treatment of ICH can reduce hematoma volume, attenuate cerebral edema and inflammation, and promote the recovery of neurological function. These findings offer a novel therapeutic strategy for ICH.

The purpose of this clinical trial is to evaluate the safety and efficacy of UC-MSCs transplantation in patients with subacute intracerebral hemorrhage, and providing a potential new therapeutic approach for this challenging condition.

DETAILED DESCRIPTION:
This clinical trial is divided into two phases: Phase I and Phase II. The Phase I clinical trial is a single-center, open-label, dose-escalation study. It follows a 3+3 dose-escalation design and includes the following phases: screening/baseline phase, stem cell treatment phase, safety and tolerability observation phase, and follow-up phase, with a total of 10 visits. The primary focus of Phase I is to assess the safety of stem cell treatment. There are three dose groups, with at least 3 subjects in each group. Each subject will receive a cell dose of 1×10^6 cells/kg, 2×10^6 cells/kg, or 4×10^6 cells/kg. Phase I will enroll patients with subacute intracerebral hemorrhage who meet all inclusion and exclusion criteria. In line with the 3+3 dose-escalation design, human umbilical cord mesenchymal stem cells (UC-MSCs) will be intravenously administered at the designated doses at specific time points. The study will then observe both the primary and secondary safety endpoints following transplantation.

The Phase II clinical trial is also a single-center, open-label study. It is an exploratory efficacy study, consisting of a screening/baseline phase, stem cell treatment phase, and follow-up phase, with 8 visits in total. The primary objective of Phase II is to evaluate the safety and efficacy of UC-MSCs in the treatment of subacute intracerebral hemorrhage. The Phase II trial will consist of two groups, each with 15 subjects, for a total of 30 participants. The specific number of cells to be transplanted will be determined based on the findings from Phase I. UC-MSCs or saline will be intravenously infused into the subjects at designated time points, and visits will be scheduled according to the study plan. The primary safety and efficacy endpoints, as well as secondary endpoints, will be closely monitored after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, gender is not limited.
2. Clinically confirmed intracerebral hemorrhage during the subacute period (3 days-10 days after onset).
3. CT confirmed as cerebral parenchymal hemorrhage, ABC/2 method to calculate the episodic hemorrhage volume of 15-30 mL (ABC/2 method hematoma volume calculation formula V (cm3) =A×B×C×1/2, A is the longest diameter of the largest level of the hematoma in the horizontal position of the CT scan (cm), B is the widest diameter of the hematoma in this plane perpendicular to the A (cm), C is the thickness of the hematoma appearing in the CT film (cm)).
4. Blood biochemical indexes meet the following conditions: 1) good coagulation function, international normalized ratio (INR) <2; 2) alachlor aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times the upper limit of the normal value, and total bilirubin <2 times the upper limit of the normal value; 3) creatinine clearance >50 mL/min; 4) hemoglobin >90 g/L; 5) absolute neutrophil value (ANC) ≥ 1.5×10^9/L, absolute lymphocyte count ≥0.4×10^9/L, platelet count ≥80×10^9/L, and albumin >25g/L; 6) procalcitonin (PCT) ≤2ng/mL.
5. National Institutes of Health Stroke Scale score (NIHSS) ≥5 and ≤20.
6. Pre-onset modified Ranking Scale score (mRS) ≤1.
7. Glasgow Coma Score (GCS) ≥9 points and ≥3 points on a single item.
8. Good compliance, signed informed consent by the person and/or legal guardian and able to receive follow-up visits at the specified time.

Exclusion Criteria:

1. Brain midline deviation >10 mm or brain hernia formation.
2. Patients who have undergone or intend to undergo surgical treatment to remove hematoma.
3. Secondary intracerebral hemorrhage caused by traumatic brain injury, arteriovenous malformation, intracranial aneurysm, coagulation disorders, hemorrhagic transformation after cerebral infarction, or tumors.
4. Suffering from malignant tumors, autoimmune diseases (including but not limited to systemic lupus erythematosus, systemic vasculitis, etc.), hemorrhagic predisposition diseases (including all kinds of hereditary hemorrhagic disorders and acquired hemorrhagic diseases), malignant cardiac arrhythmia, cardiac insufficiency (BNP ≥1000pg/mL or left ventricular ejection fraction ≤40%), acute myocardial infarction, acute or severe infectious diseases (such as intracranial infection, severe pneumonia, sepsis, etc.) and other serious diseases that may aggravate the condition and affect the assessment of efficacy.
5. Allergy or intolerance to stem cell preparations or related medicines that need to be used in the infusion process, such as saline preparations and hormone preparations.
6. Pregnant or lactating women.
7. History of stroke disease with sequelae in the last 1 year, NIHSS score ≥ 6.
8. Subarachnoid hemorrhage, primary ventricular hemorrhage, pharmacological hemorrhagic stroke.
9. Unstable vital signs, including combined respiratory abnormalities (respiratory rate <12 breaths/min or >24 breaths/min, oxygen saturation ≤90%), hyperthermia (axillary temperature >39 ℃), blood pressure ≥180/100 mmHg after antihypertensive treatment, blood glucose >20 mmol/L.
10. Those who are participating in other clinical trials.
11. Previous history of epilepsy or current use of antiepileptic drugs.
12. Unable to accept all laboratory tests and imaging tests designed by the program due to metal implants or pacemakers in the body.
13. Inability to complete the follow-up program as required.
14. Patients or their legal guardians are unwilling to sign the written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events | Up to 6 months post-transplantation
  The incidence of serious adverse events (SAEs, such as recurrent bleeding, progressive stroke, brain death, respiratory failure, renal failure, circulatory failure, secondary epilepsy, sepsis, deep vein thrombosis, etc.) and treatment-related adverse events (TEAEs, such as fever or allergies after intravenous infusion of human umbilical cord mesenchymal stem cells(UC-MSCs)) occurring within 6 months of receiving UC-MSCs therapy.
Hematoma volume | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Volume of intracerebral hemorrhage measured in cubic centimeters (cm³) as determined by quantitative analysis of head computed tomography scans.
Peri-hematomal edema volume | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Volume of edema surrounding the hematoma measured in cubic centimeters (cm³) as determined by quantitative analysis of head magnetic resonance imaging scans.
National Institutes of Health Stroke Scale (NIHSS) score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The NIHSS is a neurological examination scale that provides a quantitative measure of stroke-related neurologic deficit. Scores range from 0 to 42 points, with higher scores indicating more severe neurological impairment.
The modified Rankin Scale (mRS) score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The mRS measures the degree of disability or dependence in daily activities among individuals who have suffered a stroke. Scores range from 0 (no symptoms) to 6 (death), with higher scores indicating greater disability.
Barthel Index scale score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The Barthel Index assesses functional independence in activities of daily living across 10 items. Total scores range from 0 to 100, with higher scores indicating greater independence in activities of daily living.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 months post-transplantation
  The incidence of all non-serious adverse events occurring from infusion date through end of follow-up, including stress ulcers, pneumonia, injection site infections, and fever.
Pulmonary Embolism | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 3 weeks, 6 months post-transplantation for phase Ⅱ.
  Binary assessment (present/absent) of pulmonary embolism based on chest computed tomography with contrast enhancement.
Electrocardiogram ST Segment Deviation | Baseline and 1 day, 2 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Measurement of ST segment elevation or depression in millimeters from baseline. ST elevation ≥1mm in two or more contiguous leads or ST depression ≥0.5mm will be classified as abnormal.
Electrocardiogram Pathological Q Waves | Baseline and 1 day, 2 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Assessment for presence of pathological Q waves, defined as Q waves ≥40ms in duration or ≥25% of the height of the following R wave in at least two contiguous leads.
Electrocardiogram QTc Prolongation | Baseline and 1 day, 2 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Measurement of corrected QT interval in milliseconds. QTc intervals >450ms in males or >460ms in females will be classified as prolonged, indicating abnormal ventricular repolarization.
Electrocardiogram Arrhythmia Assessment | Baseline and 1 day, 2 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Identification and quantification of cardiac arrhythmias including atrial fibrillation, atrial flutter, ventricular tachycardia, ventricular fibrillation, and heart blocks. Results will be reported as presence or absence of each arrhythmia type.
Mini-Mental State Examination (MMSE) Score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The MMSE is a 30-point questionnaire used to measure cognitive impairment. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Montreal Cognitive Assessment (MoCA) Score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The MoCA is a cognitive screening test designed to detect mild cognitive impairment. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Hamilton Anxiety Scale (HAMA) Score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The HAMA is a 14-item scale that measures the severity of anxiety symptoms. Scores range from 0 to 56, with higher scores indicating more severe anxiety.
Hamilton Depression Scale (HAMD) Score | Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 3 months, 6 months post-transplantation for phase Ⅱ.
  The HAMD is a 17-item scale that measures the severity of depression symptoms. Scores range from 0 to 52, with higher scores indicating more severe depression.
Serum Tumor Necrosis Factor-Alpha (TNF-alpha) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of TNF-alpha in pg/mL measured in serum samples.
Serum Interleukin-1 Beta (IL-1beta) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of IL-1beta in pg/mL measured in serum samples.
Serum Interleukin-2 Receptor (IL-2R) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of IL-2R in pg/mL measured in serum samples.
Serum Interleukin-6 (IL-6) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of IL-6 in pg/mL measured in serum samples.
Serum Interleukin-8 (IL-8) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of IL-8 in pg/mL measured in serum samples.
Serum Interleukin-10 (IL-10) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I.; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of IL-10 in pg/mL measured in serum samples.
Hemoglobin Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of hemoglobin in blood measured in grams per deciliter (g/dL).
White Blood Cell Count | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Number of white blood cells per microliter (cells/μL) of blood.
Platelet Count | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Number of platelets per microliter (cells/μL) of blood.
Alanine Aminotransferase (ALT) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of ALT enzyme in international units per liter (IU/L) as a measure of liver function.
Aspartate Aminotransferase (AST) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of AST enzyme in international units per liter (IU/L) as a measure of liver function.
Blood Urea Nitrogen (BUN) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of BUN in milligrams per deciliter (mg/dL) as a measure of kidney function.
Serum Creatinine Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of creatinine in milligrams per deciliter (mg/dL) as a measure of kidney function.
Urine Protein Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of protein in urine measured in milligrams per deciliter (mg/dL).
Urine Red Blood Cell Count | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Number of red blood cells per high-power field (HPF) in urine microscopy.
Fecal Occult Blood Test | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Qualitative assessment of occult blood in stool (positive or negative).
Serum Sodium Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of sodium in serum measured in millimoles per liter (mmol/L).
Serum Potassium Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of potassium in serum measured in millimoles per liter (mmol/L).
Prothrombin Time (PT) | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Time required for plasma to clot after addition of tissue factor, measured in seconds.
Activated Partial Thromboplastin Time (aPTT) | Time required for plasma to clot after activation of intrinsic pathway, measured in seconds.
  Time required for plasma to clot after activation of intrinsic pathway, measured in seconds.
Total Cholesterol Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of total cholesterol in serum measured in milligrams per deciliter (mg/dL).
High-Density Lipoprotein (HDL) Cholesterol Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of HDL cholesterol in serum measured in milligrams per deciliter (mg/dL).
Low-Density Lipoprotein (LDL) Cholesterol Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of LDL cholesterol in serum measured in milligrams per deciliter (mg/dL).
Fasting Blood Glucose Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of glucose in blood after overnight fasting, measured in milligrams per deciliter (mg/dL).
CD4+ T Lymphocyte Count | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Number of CD4+ T lymphocytes per microliter (cells/μL) of blood as a measure of immune function.
CD8+ T Lymphocyte Count | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Number of CD8+ T lymphocytes per microliter (cells/μL) of blood as a measure of immune function.
CD4+/CD8+ Ratio | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Ratio of CD4+ to CD8+ T lymphocytes as a measure of immune system balance.
High-Sensitivity C-Reactive Protein (hs-CRP) Level | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 7 days, 2 weeks, 3 weeks, 1 month, 6 months post-transplantation for phase Ⅱ.
  Concentration of hs-CRP in milligrams per liter (mg/L) as a measure of inflammation.
Middle Cerebral Artery Blood Flow Velocity | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 6 months post-transplantation for phase Ⅱ.
  Mean blood flow velocity in the middle cerebral artery measured in centimeters per second (cm/s) using transcranial Doppler ultrasonography.
Pulsatility Index | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 6 months post-transplantation for phase Ⅱ.
  Ratio of the difference between peak systolic and end-diastolic velocities to the mean velocity in cerebral arteries as measured by transcranial Doppler ultrasonography. Higher values indicate increased vascular resistance.
Carotid Artery Stenosis Percentage | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 6 months post-transplantation for phase Ⅱ.
  Degree of carotid artery stenosis expressed as percentage reduction in vessel diameter as measured by computed tomography angiography.
Electroencephalogram Delta Wave Activity | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 3 weeks , 6 months post-transplantation for phase Ⅱ.
  Quantitative measurement of delta wave (0.5-4 Hz) power in microvolts squared (μV²). Increased focal delta activity outside of sleep states indicates abnormal cerebral function.
Electroencephalogram Epileptiform Discharges | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 3 weeks , 6 months post-transplantation for phase Ⅱ.
  Quantification of epileptiform discharges (spikes, sharp waves, spike-and-wave complexes) per hour of recording. Presence of ≥1 discharge per hour will be classified as abnormal.
Electroencephalogram Background Rhythm Analysis | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 3 weeks , 6 months post-transplantation for phase Ⅱ.
  Assessment of background rhythm frequency in Hertz (Hz) and amplitude in microvolts (μV). Normal adult awake posterior dominant rhythm is 8-13 Hz (alpha rhythm). Slowing below 8 Hz will be classified as abnormal.
Corticospinal Tract Integrity | Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 6 months post-transplantation for phase Ⅱ.
  Tractography-based assessment of corticospinal tract integrity expressed as percentage of fibers preserved compared to the unaffected hemisphere. Values range from 0% to 100%, with lower percentages indicating greater tract damage.
Electroencephalogram Hemispheric Asymmetry | Quantitative comparison of power spectral density between homologous regions of both cerebral hemispheres. Asymmetry of >50% in any frequency band will be classified as abnormal.
  Baseline and 7 days, 2 weeks, 1 month, 6 months post-transplantation for phase I; Baseline and 3 weeks , 6 months post-transplantation for phase Ⅱ.

CONTACTS AND LOCATIONS:
Overall Officials: Zhouping Tang, M.D., Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moise KJ Jr. Umbilical cord stem cells. Obstet Gynecol. 2005 Dec;106(6):1393-407. doi: 10.1097/01.AOG.0000188388.84901.e4. PMID 16319269
- [Background] Li T, Xia M, Gao Y, Chen Y, Xu Y. Human umbilical cord mesenchymal stem cells: an overview of their potential in cell-based therapy. Expert Opin Biol Ther. 2015;15(9):1293-306. doi: 10.1517/14712598.2015.1051528. Epub 2015 Jun 12. PMID 26067213
- [Background] Tsang KS, Ng CPS, Zhu XL, Wong GKC, Lu G, Ahuja AT, Wong KSL, Ng HK, Poon WS. Phase I/II randomized controlled trial of autologous bone marrow-derived mesenchymal stem cell therapy for chronic stroke. World J Stem Cells. 2017 Aug 26;9(8):133-143. doi: 10.4252/wjsc.v9.i8.133. PMID 28928910
- [Background] Chang Z, Mao G, Sun L, Ao Q, Gu Y, Liu Y. Cell therapy for cerebral hemorrhage: Five year follow-up report. Exp Ther Med. 2016 Dec;12(6):3535-3540. doi: 10.3892/etm.2016.3811. Epub 2016 Oct 18. PMID 28101148
- [Background] Hu Y, Liu N, Zhang P, Pan C, Zhang Y, Tang Y, Deng H, Aimaiti M, Zhang Y, Zhou H, Wu G, Tang Z. Preclinical Studies of Stem Cell Transplantation in Intracerebral Hemorrhage: a Systemic Review and Meta-Analysis. Mol Neurobiol. 2016 Oct;53(8):5269-77. doi: 10.1007/s12035-015-9441-6. Epub 2015 Sep 26. PMID 26409481
- [Background] Gao L, Xu W, Li T, Chen J, Shao A, Yan F, Chen G. Stem Cell Therapy: A Promising Therapeutic Method for Intracerebral Hemorrhage. Cell Transplant. 2018 Dec;27(12):1809-1824. doi: 10.1177/0963689718773363. Epub 2018 Jun 5. PMID 29871521
- [Background] Gong YH, Hao SL, Wang BC. Mesenchymal Stem Cells Transplantation in Intracerebral Hemorrhage: Application and Challenges. Front Cell Neurosci. 2021 Mar 24;15:653367. doi: 10.3389/fncel.2021.653367. eCollection 2021. PMID 33841103
- [Background] Zhou JF, Xiong Y, Kang X, Pan Z, Zhu Q, Goldbrunner R, Stavrinou L, Lin S, Hu W, Zheng F, Stavrinou P. Application of stem cells and exosomes in the treatment of intracerebral hemorrhage: an update. Stem Cell Res Ther. 2022 Jun 28;13(1):281. doi: 10.1186/s13287-022-02965-2. PMID 35765072
- [Background] Yang G, Fan X, Mazhar M, Yang S, Xu H, Dechsupa N, Wang L. Mesenchymal Stem Cell Application and Its Therapeutic Mechanisms in Intracerebral Hemorrhage. Front Cell Neurosci. 2022 Jun 13;16:898497. doi: 10.3389/fncel.2022.898497. eCollection 2022. PMID 35769327
- [Background] Mishra VK, Shih HH, Parveen F, Lenzen D, Ito E, Chan TF, Ke LY. Identifying the Therapeutic Significance of Mesenchymal Stem Cells. Cells. 2020 May 6;9(5):1145. doi: 10.3390/cells9051145. PMID 32384763
- [Background] Ding DC, Shyu WC, Lin SZ. Mesenchymal stem cells. Cell Transplant. 2011;20(1):5-14. doi: 10.3727/096368910X. PMID 21396235
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Background] Puy L, Parry-Jones AR, Sandset EC, Dowlatshahi D, Ziai W, Cordonnier C. Intracerebral haemorrhage. Nat Rev Dis Primers. 2023 Mar 16;9(1):14. doi: 10.1038/s41572-023-00424-7. PMID 36928219